CLINICAL TRIAL: NCT06920225
Title: Transmeridian Travel in Elite Female Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Professor, Florida State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005528
Record Dates: First submitted 2025-03-20; First posted 2025-04-09 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Transmeridian Travel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Home (No Intervention): Participants will perform the protocol during a home series
- Away (No Time Zone Change) (No Intervention): Participants will perform the protocol during a road series in the same time zone as home.
- Away (3 h Time Zone Change, Adopt Away Schedule) (No Intervention): Participants will perform the protocol during a road series across three time zones. The team will adopt the schedule of the new time zone.
- Away (3 h Time Zone Change, Maintain Home Schedule) (Experimental): Participants will perform the protocol during a road series across three time zones. The team will maintain the schedule of their home time zone.
  Interventions: Behavioral: Maintain home-based schedule

INTERVENTIONS:
Behavioral: Maintain home-based schedule — The team will maintain their home-based time zone schedule despite being in a location that is three time zones away
  Arms: Away (3 h Time Zone Change, Maintain Home Schedule)

SUMMARY:
The study will investigate whether maintaining a home-based time zone schedule will attenuate any decrements to sleep and performance experienced following transmeridian travel in elite female athletes.

ELIGIBILITY:
Inclusion Criteria:

* Athlete on the roster of an NCAA Division 1 Team
* Has worn WHOOP device for at least 3 months

Exclusion Criteria:

* Musculoskeletal injury or cardiometabolic disease limiting participation in regular team activities
* Pre-diagnosed sleep condition that would negatively affect sleep quantity or quality

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Sleep Quantity | Daily for 5 days
  Sleep duration will be assessed via wrist-worn WHOOP bands.
Sleep Quality | Daily for 5 days
  Sleep efficiency will be assessed via wrist-worn WHOOP bands.
Resting Heart Rate (RHR) | Daily for 5 days
  RHR will be assessed in the morning via wrist-worn WHOOP bands.
Heart Rate Variability (HRV) | Daily for 5 days
  HRV will be assessed in the morning via wrist-worn WHOOP bands.
Muscular Power | Daily for 3 days
  Muscular power is assessed via countermovement jump (CMJ) testing on force plates
Muscular Strength | Daily for 3 days
  Muscular strength is assessed via handgrip dynamometry.

SECONDARY OUTCOMES:
Reaction Time | Daily for 5 days
  Assessed in the morning via a mobile application
Subjective Sleep Quality | Daily for 5 days
  Assessed in the morning via questionnaire (0-100)
Subjective Recovery | Daily for 5 days
  Assessed in the morning via questionnaire (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences & Medicine, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Some of the individual data collected on the athletes is confidential to the research team and the team(s) participating in the study.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT06920225/ICF_000.pdf